CLINICAL TRIAL: NCT05837728
Title: More Good Days At Home: Advancing Health-promoting Practices in Municipal Healthcare Services for Older Recipients of Home Care
Brief Title: Health Determinants in Older Adults Living At Home
Status: Completed | Type: Observational
Sponsor: University of Stavanger (Other)
Collaborators: Stavanger Municipality, Norway (Unknown)
Responsible Party: Sponsor
Other Study IDs: 320622
Record Dates: First submitted 2023-03-20; First posted 2023-05-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Frailty; Vision and Hearing Loss; Cognitive Function, Social 1; Mental Health Issue; Social Functioning; Alcohol Use, Unspecified; Healthy Aging
MeSH Terms: conditions — Frailty; Deaf-Blind Disorders; Social Adjustment; Alcohol Drinking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older adults ≥75 living at home: Older adults ≥75 years living at home applying for a municipal health and care service for an estimated period of more than two weeks.
  Interventions: Behavioral: Health promoting assessment of older adults living at home

INTERVENTIONS:
Behavioral: Health promoting assessment of older adults living at home — Based on the results of the first assessment of the older person's health determinants, healthcare professionals will recommend and tailor measures to the individual's needs to reduce the risk of functional decline and maintain their health while living at home.

SUMMARY:
The observational study will conduct interprofessional assessments by registered nurses, physiotherapists, and occupational therapists of health determinants (i.e., frailty, physical, cognitive, and sensory function, mental and social health, and alcohol use) in older adults (≥75) living at home and applying for a municipal health service. The participants will take part in two assessments, baseline and 5 months. Based on the baseline assessment healthcare professionals will identify factors that can affect older adults' health, provide tailored information, offer measures, and link with proper health services. The aim is that older adults maintain health, function, and self-care and thus can continue aging at home. The main research question is:) How can interprofessional assessments of older adults living at home reduce the risk of impaired function, maintain health and ensure that the elderly receive tailored services?

DETAILED DESCRIPTION:
The population of older adults is rapidly increasing worldwide and in Norway. A present and future challenge is to provide adequate health and care services to older persons. It is imperative to organize the services in a manner that is both adequate for the older persons in need of help and sustainable for health and care services and society. A way to ensure this is to facilitate and promote measures allowing older adults to age well at home. Accordingly, it is of great importance to enable older adults to engage with health determinants that influence their daily life actively. One area of importance is assessing health determinants and acting upon indications of functional decline, cognitive and sensory impairments, and frailty.

The observational study will assess how interprofessional assessments of health determinants in older adults living at home can promote health and reduce the risk of functional decline. The study participants will take part in two assessments of health determinants including frailty, physical, cognitive, and sensory function, mental and social health, and alcohol use. Based on results from the baseline assessment healthcare personnel will identify factors that can affect the older adult's health, provide tailored information to strengthen health literacy, and offer measures available in the health services in the municipality. The second assessment 5 months after baseline will reveal if tailoring measures and services have contributed to maintaining and supporting the older person's health and reduced the risk of functional decline. The aim of the project is that the elderly living at home maintains health, function, and self-care and thus can have more good days at home.

ELIGIBILITY:
Inclusion Criteria:

* Older adults, age ≥75, live at home, being cognitively able to give informed consent, apply for a public health and care service from the municipality, and have a service need for more than two weeks approved by the municipality

Exclusion Criteria:

* <75 years, cognitive impairment, in need of palliative services

Ages: 75 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Home-living older adults applying for municipal health services.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Measure of Physical function | Baseline and 5 Months
  Change in the older adult's physical function will be measured with the "Short Physical Performance Battery". Values: 0-4. A higher score means better physical function.
Measure of cognitive function | Baseline and 5 Months
  Change in the older adult's cognitive function will be measured with the "MiniCog" screening tool for cognitive impairment.
  Values: 0-4. We use a cut-off value of <4 points which is recommended, as this may indicate a need for further investigation of cognitive status.
Measure of clinical frailty | Baseline and 5 Months
  Change in frailty will be measured with the "Global Measure of frailty and fitness in elderly people".
  Values: 0-9. A higher score means a high level of frailty.
Measure of lonliness | Baseline and 5 Months
  Change in lonliness will be measured with "The Short UCLA Lonliness scale". Values: 0-3. A higher score means a high level of lonliness.
Measure of depression | Baseline and 5 Months
  To assess change in depression in old age, we will use the 4-item Geriatric Depression Scale (GDS).Values: 0-1. A cut-off score >0 indicates depression
Measure of alcohol use | Baseline and 5 Months
  For assessment of change in alcohol consumption, we will use the Alcohol Use Disorders Identification Test (AUDIT-C) 4 items. Values:0-12.The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the person's drinking is affecting his/her health.
Measure of vision | Baseline and 5 Months
  Change in vision will be measured with a structured vision assessment tool called KROSS (a Norwegian acronym for Competence, Rehabilitation of Sight after Stroke) developed by the University of South-Eastern Norway in collaboration with the Vestre Viken Hospital Trust and stroke survivor organizations. The KROSS tool includes assessments of visual acuity, visual field, eye alignment and movements, and visual attention.
Measure of hearing | Baseline and 5 Months
  Change in hearing will be measured with the Combined Serious Sensory Impairment (Kombinert Alvorlig Sansesvikt) KAS- Screen interview guide. The questions used in our study come from the hearing and verbal communication/social life subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Storm, PhD, Principal Investigator — Universitetet i Stavanger; Grethe Eilertsen, PhD, Principal Investigator — University of South-Eastern Norway
Locations (1):
- Stavanger kommune, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kvalsvik F, Larsen BH, Eilertsen G, Falkenberg HK, Dalen I, Haaland S, Storm M. Health Needs Assessment in Home-Living Older Adults: Protocol for a Pre-Post Study. JMIR Res Protoc. 2024 Apr 18;13:e55192. doi: 10.2196/55192. PMID 38635319